CLINICAL TRIAL: NCT01021917
Title: Weight Loss & Maintenance of Weight Loss Tracking Study (SUCCESS Tracking Study)
Brief Title: SUCCESS Tracking Study
Status: Terminated | Type: Observational
Why Stopped: Given the length of time data was collected (i.e. 5 1/3 years), we do not anticipate a change any potential conclusions by completing the final survey.
Sponsor: Medifast, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MED013; 20071961 (Other: Western Institutional Review Board)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Meal Replacements
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Other Dieters (OD): Those participating in weight loss programs other than Medifast Direct or Take Shape For Life.
- Take Shape For Life (TSFL): Those using Medifast meal replacement products for weight loss while working closely with a Take Shape For Life certified Health Coach.
- Medifast Direct (MD): Those using Medifast meal replacement products specifically for weight loss that were purchased directly from the company and individually monitored by the customer.

SUMMARY:
The overall purpose of this research is to evaluate the long-term outcomes associated with participation in Medifast Direct and Take Shape For Life weight-loss programs in comparison with non-Medifast weight-loss programs. Another important goal of this research is to determine whether the differences between Medifast Direct and Take Shape For Life programs affect weight-loss and maintenance of weight-loss in customers.

DETAILED DESCRIPTION:
Researchers desire to capture the behaviors and outcomes of those individuals who would enroll in these programs without the additional encouragement to be a participant in a research study. The study will employ an observational prospective design intended to introduce as little interference as possible with subjects' behaviors. This is in order to capture the pure effects of the weight-loss programs themselves, and to reduce the potentially confounding effects of merely participating in a research study. Subjects who have already committed to a weight-loss program (Medifast Direct, Take Shape For Life , or other) will be recruited to join this study, and will be asked to complete several questionnaires over a period of up to 6 ⅓ years after enrollment. Questionnaires will measure information regarding anthropometrics, sociodemographics, and health & quality of life outcomes. The overall goal of this research is to be able to describe and compare the long-term dieting behaviors and outcomes among participants in Medifast Direct and Take Shape For Life programs in comparison with other dieters.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females between the ages of 18 - 69 years
* BMI ( > 25.0 kg/m2)
* Beginning a weight loss diet plan (MD, TSFL, or one of a number of commercially available plans)NOTE: subjects must have already committed to a weight-loss plan in order to be eligible for this study. The recruitment process is specifically designed so as NOT to appear to encourage subjects to begin a weight-loss plan. Rather, the purpose of this research is to track information about persons who have already committed to a weight-loss program.
* Willing and able to give informed consent
* Willing and able to comply with study protocol

Exclusion Criteria:

* Unable to give informed consent
* Previous hospitalization for psychiatric disorder or eating disorder
* Current, uncontrolled medical conditions
* Taking unstable doses of weight-loss or appetite-affecting medications (e.g., SSRIs, steroids, Ritalin)
* Taking prescription weight-loss drugs (Phentermine, Sibutramine, Orlistat, etc…)
* Have undergone, or plan to undergo, weight loss surgery (e.g. gastric bypass, lap band, duodenal switch) in the next 6 1/3 years
* Plan to undergo weight-altering cosmetic surgery procedures (e.g. breast reduction/augmentation, tummy tuck, liposuction, or other skin removal procedures) in the next 6 1/3 years

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To compare change in body weight among subjects in Medifast Direct, Take Shape For Life, and Other Dieters. | 4 months, 16 months, and at 5y follow-up

SECONDARY OUTCOMES:
To investigate attrition rates among subjects enrolled in Medifast Direct, Take Shape For Life, and Other Dieters. | 4 months, 16 months, and at 5 yr follow-up
To evaluate potential predictors of successful weight loss & maintenance of weight loss. | 4 months, 16 months, and at 5 yr follow-up
To examine the effects of Medifast Direct and Take Shape For Life programs on intake, health & quality of life outcomes, and eating behaviors. | 4 months, 16 months, and at 5y follow-up
To explore potential differences between subgroups in change in body weight and attrition. | 4 months, 16 months, and at 5y follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Davis, PhD, Principal Investigator — Medifast, Inc.; Christopher D Coleman, MS, Study Director — Medifast, Inc.
Locations (1):
- Medifast Inc., Owings Mills, Maryland, United States

REFERENCES:
- [Background] Thearle M, Aronne LJ. Obesity and pharmacologic therapy. Endocrinol Metab Clin North Am. 2003 Dec;32(4):1005-24. doi: 10.1016/s0889-8529(03)00066-5. PMID 14711072
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Gale SM, Castracane VD, Mantzoros CS. Energy homeostasis, obesity and eating disorders: recent advances in endocrinology. J Nutr. 2004 Feb;134(2):295-8. doi: 10.1093/jn/134.2.295. PMID 14747663
- [Background] Heymsfield SB, van Mierlo CA, van der Knaap HC, Heo M, Frier HI. Weight management using a meal replacement strategy: meta and pooling analysis from six studies. Int J Obes Relat Metab Disord. 2003 May;27(5):537-49. doi: 10.1038/sj.ijo.0802258. PMID 12704397
- [Background] Ditschuneit HH, Flechtner-Mors M, Johnson TD, Adler G. Metabolic and weight-loss effects of a long-term dietary intervention in obese patients. Am J Clin Nutr. 1999 Feb;69(2):198-204. doi: 10.1093/ajcn/69.2.198. PMID 9989680
- [Background] Ditschuneit HH, Flechtner-Mors M. Value of structured meals for weight management: risk factors and long-term weight maintenance. Obes Res. 2001 Nov;9 Suppl 4:284S-289S. doi: 10.1038/oby.2001.132. PMID 11707555
- [Background] Quinn Rothacker D. Five-year self-management of weight using meal replacements: comparison with matched controls in rural Wisconsin. Nutrition. 2000 May;16(5):344-8. doi: 10.1016/s0899-9007(99)00280-4. PMID 10793302
- [Background] Glenny AM, O'Meara S, Melville A, Sheldon TA, Wilson C. The treatment and prevention of obesity: a systematic review of the literature. Int J Obes Relat Metab Disord. 1997 Sep;21(9):715-37. doi: 10.1038/sj.ijo.0800495. PMID 9376884
- [Background] Golan M, Weizman A, Apter A, Fainaru M. Parents as the exclusive agents of change in the treatment of childhood obesity. Am J Clin Nutr. 1998 Jun;67(6):1130-5. doi: 10.1093/ajcn/67.6.1130. PMID 9625084
- [Background] Stata Statistical Software: release 7.0 College Station TX. Stata Corporation: College Station, TX 1994-2001.